CLINICAL TRIAL: NCT06604455
Title: Impact of Acupuncture and Integrative Medicine on Patients' Quality-of-life During National Emergency and Wartime in Integrative Oncology and Inpatient Settings
Brief Title: Impact of Acupuncture and Integrative Medicine on Patients Quality-of-life During National Emergency and Wartime
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Eran Ben-Arye, Director, Integrative Oncology Program, Carmel Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CMC-24-0046
Record Dates: First submitted 2024-09-17; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Supportive Care
Keywords: Integrative medicine; Integrative oncology; acupuncture
MeSH Terms: interventions — Acupressure; Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Integrative medicine single-modality (Experimental): Acupressure/relaxation only
  Interventions: Other: acupressure/relaxation
- Integrative medicine multi-modality (Experimental): Acupressure/relaxation with acupuncture
  Interventions: Other: acupressure/relaxation with acupuncture

INTERVENTIONS:
Other: acupressure/relaxation with acupuncture — The acupressure/acupuncture points will be designated based on evidence-based research. For example, clinical guideline-based integrative oncology protocol for pain relief will include the following analgesia-related acupressure/acupuncture points: Liver-3, Taichong; Large-Intestine 4, Hegu; Stomach-36, Zusanli; Pericard-6, Neiguan; Spleen-6, Sanyinjiao; Yin tang; as well as battlefield ear acupuncture points. In both intervention groups, relaxation techniques will be tailored to the patient's quality of life related concerns, with the option of including breathing and guided imagery modalities as well.
  Arms: Integrative medicine multi-modality
Other: acupressure/relaxation — The acupressure points will be designated based on evidence-based research. In both intervention groups, relaxation techniques will be tailored to the patient's quality of life related concerns, with the option of including breathing and guided imagery modalities as well.
  Arms: Integrative medicine single-modality

SUMMARY:
The current ongoing war in Israel, which began in October 2023 with a risk for spreading regionally across the Middle East, has presented a significant challenge to many patients, affecting also those receiving active oncology treatment. The present study examines a unique setting of care involving a diverse population of patients, including those receiving oncology treatment, from a widely diverse social, cultural and religious, background. Patients are offered integrative medicine treatments for 3 weeks with the goal of addressing war-related physical, emotional, and other quality of life-related concerns. After signing the informed consent form, patients will be randomly allocated to one of the two study interventions: acupressure-relaxation alone (Group A); or acupressure-relaxation modalities with acupuncture (Group B). The response to the study intervention for quality of life-related concerns will be re-assessed immediately; at 24-48 hours; and after 3 weeks following the treatment. Patients will also undergo objective measurements during treatment using Heart Rate Variability (HRV) to determine the impact of the intervention on their QoL and concerns.

DETAILED DESCRIPTION:
Integrative medicine is increasingly being included in supportive and palliative care, primarily in oncology settings. The current military conflict in Israel has led to a surge in cases of emotional and physical distress, overwhelming the health profession throughout the country.

Study objectives and purpose: The primary study objective is to improve patients' QoL-related concerns including those affected by the military conflict.

Study design and setting: The study is taken place within a prospective randomized controlled methodology.

Study population: Patients of either gender, hospitalized for various indications (oncology or not) or undergoing out-patient oncology treatment, age ≥ 18 years.

Allocation to study arms and groups: Participants will be randomly assigned using the "Research Randomizer" online tool (https://www.randomizer.org/) to one of the following study groups:

* Single-modality integrative medicine, receiving acupressure/relaxation only (Group A)
* Multi-modality integrative medicine receiving acupressure/relaxation with acupuncture (Group B) In both study groups, the interviews will address quality of life-related concerns, including war-related concerns. Reassessment of these concerns will be conducted immediately post-treatment, 24-hour post treatment and following 3 weeks. patients in both groups will be offered weekly integrative medicine treatments during the 3 weeks following the first treatment .

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with cancer, age ≥ 18 years who are either hospitalized or undergoing oncology treatment in an outpatient care setting; or hospitalized for any other diagnosis
* Patients expressing quality of life related concerns affected directly or indirectly to the war and related security status.

Exclusion Criteria:

Inability to read and provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-08-28 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Assessing patients' quality of life-related concerns using the Measure Yourself Concerns and Wellbeing (MYCAW) | Before and immediately following the integrative medicine intervention; at 24-48 hours; and three weeks post-treatment.
  In MYCAW, patients are asked to list and then score (from 0 to 6; 6 is most severe) their 2 most severe quality of life-related concerns
Assessment of objective physiological changes during the intervention | During the 30 minutes integrative medicine intervention
  Assessment of objective physiological changes during the 30-minute integrative medicine intervention will be conducted using chest-lead electrocardiogram monitoring autonomic heart rate variability (HRV) throughout.

SECONDARY OUTCOMES:
Assessing patients' QoL-related concerns using the Edmonton Symptom Assessment Scale (ESAS) | Before and immediately following the integrative medicine intervention; at 24-48 hours; and three weeks post-treatment.
  ESAS asks respondents to score a list of 10 QoL-related concerns on a scale from 0 (no symptom) to 10 (worst severity of the symptom).
Assessing patients' quality of life-related concerns using the European Organization for Research and Treatment of Cancer Quality of Life (EORTC QLQ-C30) | Before and three weeks post-treatment.
  EORTC QLQ C-30 asks a number of quality of life-related clusters of concerns, from 1 (not at all) to 4 (very much).

CONTACTS AND LOCATIONS:
Overall Officials: Eran Ben-Arye, MD, Principal Investigator — Director, Integrative Oncology Program
Locations (1):
- Carmel Medical center, Haifa, Israel, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sowan W, Baziliansky S. Acute Stress Symptoms, Intolerance of Uncertainty and Coping Strategies in Reaction to the October 7 War. Clin Psychol Psychother. 2024 May-Jun;31(3):e3021. doi: 10.1002/cpp.3021. PMID 38894501